CLINICAL TRIAL: NCT06059508
Title: A Multicenter, Open-label Phase I Clinical Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of SHR-5495 for Injection in Patients With Advanced Malignancies
Brief Title: Phase I Clinical Study of SHR-5495 in the Treatment of Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-5495-I-101
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-07

CONDITIONS: Advanced Malignant Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-5495 for injection (Experimental)
  Interventions: Drug: SHR-5495 for injection

INTERVENTIONS:
Drug: SHR-5495 for injection — SHR-5495 for injection

SUMMARY:
This study is an open, multicenter, dose-increasing/dose-expanding/efficacy expanding Phase I clinical study aimed at evaluating the tolerance, safety, PK, PD, and immunogenicity of SHR-5495 in the treatment of advanced malignant tumor patients, and preliminarily observing its anti-tumor efficacy. The entire study was divided into three stages: dose escalation, dose extension, and efficacy extension.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 70 years old (including 18 and 70 years old), both male and female
2. Pathologically confirmed advanced malignant tumors that have failed sufficient standard treatment or have no effective standard treatment plan
3. ECOG score: 0-1
4. Expected survival time ≥ 12 weeks
5. Existence of measurable lesions that meet RECIST 1.1 standards
6. Sufficient Hematology and end organ function shall be completed within 7 days before the first study treatment
7. Left ventricular Ejection fraction (LVEF) ≥ 50% within 28 days before the first administration
8. Women of childbearing age must carry out serum Pregnancy test within 7 days before the first administration, and the result is negative. Female subjects of childbearing age and male subjects with partners of childbearing age must agree to use efficient methods of contraception or abstinence within at least 26 weeks (female subjects) or 14 weeks (male subjects) from the date of signing the informed consent form until the last administration
9. The patient voluntarily joined this study, signed an informed consent form, had good understand the research procedures, and have signed informed consent

Exclusion Criteria:

1. Has received treatment with interleukin
2. Previously received immune checkpoint inhibitors
3. Central nervous system metastasis with clinical symptoms in patients
4. The third space effusion with clinical symptoms needs repeated drainage, such as pericardial effusion, Pleural effusion and peritoneal effusion that cannot be controlled after pumping or other treatment
5. Subjects who received anti-tumor therapy and systemic immune stimulation therapy within 4 weeks prior to the first dose of the study drug; Received traditional Chinese patent medicines and simple preparations anti-tumor treatment within 2 weeks before the first dose of study drug
6. Subjects who received>30Gy of non thoracic radical radiation therapy within 28 days before the first medication, those who received>30Gy of chest radiation therapy within 24 weeks before the first medication, and those who received ≤ 30Gy of palliative radiation therapy within 14 days before the first medication
7. Subjects who have received systemic Immunosuppressive drug treatment within 2 weeks before the first administration, or who are expected to require systemic immunosuppressive drug treatment during the study treatment.
8. Patients who have not recovered to ≤ CTCAE level 1 (CTCAE v5.0) due to adverse events caused by previous treatment
9. Having autoimmune diseases
10. Other malignant tumors within 2 years before screening, excluding fully treated cervical Carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal Carcinoma in situ after radical surgery
11. Subjects with known or suspected interstitial pneumonia; Other moderate to severe lung diseases that may interfere with the detection or treatment of drug-related pulmonary toxicity and seriously affect respiratory function
12. Subjects with severe cardio cerebral Vascular disease
13. Clinically significant bleeding symptoms or tendency to bleed within one month before the first administration
14. Arteriovenous thrombotic events that occurred within 3 months before the first administration
15. Uncontrolled tumor related pain or symptomatic hypercalcemia. Subjects who require painkillers must already have a stable painkillers treatment plan at the time of entry into the study; Symptomatic lesions suitable for palliative radiotherapy should be treated before entering the study
16. Active hepatitis B or active hepatitis C
17. Abnormal electrocardiogram (ECG) examination, judged by the researcher to have clinical significance
18. Have a history of immune deficiency
19. Evidence of active tuberculosis infection within 1 year prior to the first administration, or a history of active tuberculosis infection more than 1 year ago without formal treatment
20. Serious infection occurred within 4 weeks before the first administration; Active infections that have received therapeutic intravenous or oral antibiotics within 2 weeks prior to starting the study.
21. History of live attenuated vaccine administration within 28 days prior to initial administration or expected study period
22. Within 28 days prior to the first administration, major surgeries other than diagnosis or biopsy have been performed; Traumatic minor surgery experienced within 7 days prior to first administration
23. Subjects who have previously received or are preparing to receive allogeneic bone marrow transplantation or solid organ transplantation
24. Has a history of severe allergic reactions to other monoclonal antibodies/fusion protein drugs, and is allergic to any component of the research treatment plan
25. Female subjects during pregnancy, lactation, or planning to conceive during the study period
26. The subject has a known history of psychotropic substance abuse, alcoholism, or drug abuse
27. Researchers believe that any other medical, psychiatric, or social condition may interfere with the subjects' rights, safety, health, or ability to sign informed consent, cooperate and participate in the study, or interfere with the evaluation of the study medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) of SHR-5495 | up to 21 days
AEs+SAEs | from the first drug administration to within 90 days for the last treatment dose
Maximum tolerated dose（MTD）of SHR-5495 | up to 21 days
Maximum administrated dose（MAD）of SHR-5495 | up to 21 days
Recommended Phase II Dose (RP2D) of SHR-5495 | up to 21 days

SECONDARY OUTCOMES:
Evaluation of pharmacokinetic parameter of SHR-5495: Cmax | 12 months
Evaluation of pharmacokinetic parameter of SHR-5495: Tmax | 12 months
Evaluation of pharmacokinetic parameter of SHR-5495: AUClast | 12 months
Evaluation of pharmacokinetic parameter of SHR-5495: AUCinf | 12 months
Evaluation of pharmacokinetic parameter of SHR-5495: t1/2 | 12 months
Evaluation of pharmacokinetic parameter of SHR-5495: CL | 12 months
Evaluation of pharmacokinetic parameter of SHR-5495: Vss | 12 months
Receptor occupancy rate | 12 months
Objective Response Rate (ORR) | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Duration of response (DoR) | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Disease control rate (DCR) | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Progression free survival（PFS） | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Overall survival (OS) | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Target cell count | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong First Medical University Affiliated Cancer Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided